CLINICAL TRIAL: NCT03608137
Title: Cannabis and Thought Disorder in Schizophrenia: Clinical and Neuroimaging Relationships
Brief Title: Cannabis and Thought Disorder in Schizophrenia
Acronym: CANDI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminée
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A00062-53
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia ; Cannabis
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis users (Experimental): Subjects of this group have to meet the DSM-5 criteria for schizophrenia and smoke cannabis at least two days per week for every week of the past month. They have to exhibit negative urine screen for any substance except benzodiazepines and cannabis.
  Interventions: Other: Cannabis and thought disorder in schizophrenia:clinical and neuroimaging relationships
- Non- cannabis users (control group) (Active Comparator): Subjects of this group have to meet the DSM-5 criteria for schizophrenia and have to report no cannabis use over the previous month, and exhibit negative urine screen for any substance except benzodiazepines.
  Interventions: Other: Cannabis and thought disorder in schizophrenia:clinical and neuroimaging relationships

INTERVENTIONS:
Other: Cannabis and thought disorder in schizophrenia:clinical and neuroimaging relationships — To investigate whether the level of cannabis use in schizophrenic patients influences the symptoms of psychic disorganization via modulation of cerebral connectivity between the temporal lobe and the putamen.

SUMMARY:
Recent studies have suggested a strong relationship between cannabis use and the level of thought disorder in subjects with schizophrenia. Moreover, the level of thought disorder has been associated with an increased functional connectivity between the temporal lobe and the Putamen. However, the brain mechanisms underlying these two relationships are still poorly known. Better understanding these mechanisms is important to improve patients' care, in particular among treatment-resistant patients.

The objective of the CANDI study consists of assessing whether the level of cannabis use in patients with schizophrenia modulates the level of thought disorder via a modulation of the functional connectivity between the temporal lobe and the Putamen. Analyses will be controlled for the composition of cannabis, in particular the tetrahydrocannabinol / cannabidiol ratio.

DETAILED DESCRIPTION:
25 subjects with schizophrenia and current cannabis use will be recruited in the experimental group. The control group will consist of 25 subjects with schizophrenia but with no cannabis use.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Meeting the DSM-5 criteria for schizophrenia
* "Cannabis user" group: - Smoking at least two days per week during the previous months
* Displaying positive urine screen for cannabis
* "Non-cannabis user" group: - No episode of cannabis smoking during the previous month
* Negative urine screen for cannabis + no lifetime criteria for cannabis use disorder (assessment by an addiction specialist).

Exclusion Criteria:

* Current criteria for axis-1 psychiatric disorder other than schizophrenia
* Current criteria for any other substance use disorder except for nicotine use disorder
* Any contraindication for MRI
* Tutorship or curatorship
* Pregnant or lactating woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Level of thought disorder | one year
  The level of thought disorder will be investigated using the specific items of the Positive And Negative Syndrome Scale (PANSS; Kay et al., 1987) Minimum score 1 Maximum score 7

SECONDARY OUTCOMES:
cannabis use | one year
  cannabis use (yes vs. no; i.e., the group factor)
Delta-9 tetrahydrocannabinol (THC) concentration | one year
  Concentrations of Delta-9 tetrahydrocannabinol in the cannabis usually smoked
Cannabidiol (CBD) concentration | one year
  Concentration of cannabidiol in the cannabis usually smoked

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, MD, PhD, Principal Investigator — CH LE VINATIER; Guillaume SESCOUSSE, MD, Study Director — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No